CLINICAL TRIAL: NCT06144541
Title: Correlation Between Objective Skin Pigment Measurement and Fitzpatrick Skin Type
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Responsible Party: Sponsor
Other Study IDs: i23-09_Fitz_Skin
Record Dates: First submitted 2023-10-12; First posted 2023-11-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Skin Pigment
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General public: This survey and ITA measurements will be performed among the general public
  Interventions: Other: Survey administration for Fitzpatrick skin type; Device: Measurement of ITA based on SkinColorCatch instrument

INTERVENTIONS:
Other: Survey administration for Fitzpatrick skin type — Survey administration for Fitzpatrick skin type
Device: Measurement of ITA based on SkinColorCatch instrument — Measurement of ITA based on SkinColorCatch instrument

SUMMARY:
The purpose of this study is to correlate subjective skin pigment measurements as reported by patient-responses to the Fitzpatrick Skin Type Scale versus objective classification of skin pigment utilizing Individual Typology Angle (ITA) measurements.

DETAILED DESCRIPTION:
The Fitzpatrick scale is a numerical classification for human skin color developed in 1975 as a way to estimate the response of different types of skin to UV light. It is used by dermatologists to classify skin tone and assess the risk of skin cancer.

The Fitzpatrick scale encompasses six gradings, from I to VI. However, this does not include all skin tones, as there are significantly more not encompassed within the scale. The aim of this study is to incorporate objective measurements when identifying a patient's Fitzpatrick skin type.

ELIGIBILITY:
Inclusion Criteria:

* Male and females that are 18 years of age and older
* Subjects with all Fitzpatrick skin types I-VI One-third of subjects will be Fitzpatrick I or II skin types, one-third of subjects will be III or IV, and one-third will have V and VI.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners
* Adults unable to consent
* Individuals with open wounds on the nondominant upper inner arm
* Individuals with fibrotic skin disease or other skin conditions or hair growth on the nondominant upper inner arm that could affect skin measurements in the opinion of the investigator
* Individuals with tattoos that cover the site on the nondominant upper inner arm
* Individuals with post-inflammatory hypopigmentation or hyperpigmentation
* Individuals with vitiligo
* Individuals who have used self-tanning products or tanning beds in the last two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects, healthy and unhealthy, are eligible to enroll. Subjects from the greater Sacramento region will be enrolled. Subjects must be at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Skin colorimeter derived Individual Typology Angle value correlated against self-reported Fitzpatrick skin type | One time - collected for up to 1 year for the entire study
  Correlation of ITA by the use of SkinColorCatch (Delfin) compared to the Fitzpatrick skin scale as determined by the patients' responses to validated questionnaire.
  The higher the ITA, the lighter the skin. ITA skin color types are classified into six groups, from Very Light to Dark skin.

SECONDARY OUTCOMES:
Assess Fitzpatrick Skin type based on validated questionnaire | One time - collected for up to 1 year for the entire study
  Questionnaire about sun sensitivity and tanning will be administered to calculate the Fitzpatrick skin types
Sun protection habit use | One time - collected for up to 1 year for the entire study
  Quantification of sun protection habits based on survey question asking their typical use of sun protection

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science & Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No